CLINICAL TRIAL: NCT06658938
Title: A Prospective, Single-arm Clinical Study of Blinatumomab in the Maintenance Treatment of High-risk Patients With Acute B-lymphoblastic Leukemia After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Blinatumomab as Maintenance Therapy in Patients With High-risk B-lineage Acute Lymphoblastic Leukemia Post Allogeneic Hematopoietic Cell Transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024066
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-09

CONDITIONS: B-ALL
Keywords: allogeneic hematopoietic stem cell transplantation
MeSH Terms: interventions — blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with B-ALL receiving allogeneic hematopoietic stem cell transplantation (Other)
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Beginning 3 months after transplantation, 1 cycle of blinatumomab was performed every 3 months for a total of 4 maintenance cycles.
  Dosage of blinatumomab: 9 ug/d D1-4, 28 ug/d D5-14

SUMMARY:
Patients ≥ 14 years of age after B-ALL allogeneic transplantation received 4 cycles of maintenance therapy with blinatumomab +/- TKI and were followed for more than 1 year to assess overall survival (OS), relapse-free survival (RFS), incidence of acute and chronic GVHD, safety, etc.

DETAILED DESCRIPTION:
Patients ≥ 14 years of age after B-ALL allogeneic transplantation received 4 cycles of maintenance therapy with blinatumomab +/- TKI and were followed for more than 1 year to assess overall survival (OS), relapse-free survival (RFS), incidence of acute and chronic GVHD, safety, etc.

Beginning 3 months after transplantation, 1 cycle of blinatumomab was performed every 3 months for a total of 4 maintenance cycles.

Dosage of blinatumomab: 9 ug/d D1-4, 28 ug/d D5-14

ELIGIBILITY:
Inclusion Criteria:

* 1．Age ≥ 14 years, male or female; 2．CD19 + acute B lymphoblastic leukemia treated with allogeneic hematopoietic stem cell transplantation [Patients, the types of transplantation include fully matched sibling transplantation, haploidentical related donor transplantation and unrelated donor transplantation; 3．CD19 + acute B-lymphoblastic leukemia at risk of relapse before transplantation [including but not limited to: refractory leukemia: failure to achieve complete remission (CR)/CR with partial hematological recovery (CRh)/CR with incomplete hematological recovery (CRi) or CR/CRh/CRi after the end of induction therapy (generally refers to 4-week regimen or Hyper-CVAD regimen), but still positive for measurable residual disease (MRD); relapsed leukemia: patients who have achieved CR have blasts in peripheral blood or bone marrow (proportion > 5%), or extramedullary disease; onset of white blood cells > 30 × 109/L; patients with poor prognosis cytogenetic abnormalities; patients with positive residual leukemia before transplantation, etc.] 4．The disease is in complete remission, and residual leukemia is negative, absolute neutrophil count ≥ 1.0 × 109/L, platelet count ≥ 50 × 109/L, lasting for more than a week; 5．Freedom from ≥ Grade 3 acute GVHD or uncontrolled moderate to severe chronic GVHD within 30 days prior to enrollment; Awareness and willingness to sign written informed consent.

Exclusion Criteria:

* 1.Patients with hematological relapse or minimal residual disease relapse of B-ALL after transplantation; 2.Presence of serious uncontrolled active infection (e.g., sepsis, pulmonary infection, etc.).

  3.Markedly abnormal screening laboratory tests: A) Alanine aminotransferase (ALT) ≥ 5 × ULN (upper limit of normal); B) Aspartate aminotransferase (AST) ≥ 5 × ULN; C) Total bilirubin (TBIL) ≥ 3 × ULN; D) Creatinine clearance < 70 mL/min at screening; Patients with active hepatitis B (hepatitis B surface antigen positive and peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) ≥ 1 × 102 copies/mL); F) Hepatitis C antibody positive; G) Human immunodeficiency virus (HIV) positive; h) Treponema pallidum antibody positive; 4.ECOG performance status ≥ 3 5.Estimated survival less than 3 months This study may not be completed for other reasons, or the investigator considers it inappropriate to participate in this study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
CIR) | 2 years
  Cumulative recurrence rate (CIR)

SECONDARY OUTCOMES:
OS | 2 years
  2 Overall survival (OS)
RFS | 2 years
  relapse-free survival (RFS)
incidence of acute and chronic GVHD | 1-year
  incidence of acute and chronic GVHD